CLINICAL TRIAL: NCT02420392
Title: Effects of Dapagliflozin on the Incretin Sensitivity of the Pancreatic Beta Cell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Young Min Cho, Assistant Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H1407-176-598
Record Dates: First submitted 2015-04-11; First posted 2015-04-17 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapagliflozin treatment (Experimental): Test incretin sensitivity after dapagliflozin treatment in type 2 diabetes patients
  Interventions: Drug: Dapagliflozin
- Normal glucose tolerance (No Intervention): Test incretin sensitivity in subjects with normal glucose tolerance

INTERVENTIONS:
Drug: Dapagliflozin — 8 weeks treatment of dapagliflozin added to the type 2 diabetes patients with unsufficiently controlled with metformin or sulfonylurea
  Arms: Dapagliflozin treatment

SUMMARY:
To investigate the effect of dapagliflozin on the incretin sensitivity of the pancreatic beta cell.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for dapagliflozin arm
* Normal glucose tolerance (fasting plasma glucose <100 mgd/l, HbA1c <6.0%) for normal glucose tolerance arm
* Age 18 to 75 years
* BMI <35 kg/m2
* For type 2 diabetes patients, at least 3 months of treatment period and HbA1c 7.5 to 11.0% and treatment with lifestyle modification and/or metformin or sulfonylurea

Exclusion Criteria:

* Who is allergic to dapagliflozin
* Type 1 diabetes
* Patients with history of diabetic ketoacidosis
* Reduced renal function (eGFR <60ml/min/1.73m2)
* Taking loop diuretics or dehydrated patient
* History of hypotension when taking hypertensive medication
* Diagnosed with heart failure
* Diagnosed with cerebral infarction
* Taking insulin, DPP-4 inhibitor, GLP-1 analogue, pioglitazone, alpha-glucosidase inhibitor
* Above upper limit of normal hematocrit range (male 39-52%, female 36-48%)
* Pregnant or breastfeeding women
* History of recurrent genitourinary infection
* AST/ALT more than two fold increased above normal upper limit
* Hemolytic disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Difference of incretin sensitivity of pancreatic beta cell measured by hyperglycemic clamp with GLP-1 and GIP infusion | From 60 minutes to 120 minutes during GLP-1 infusion under hyperglycemic clamp
  Area under the curve of C-peptide level during GLP-1 infusion under hyperglycemic clamp

SECONDARY OUTCOMES:
First phase insulin/C-peptide response | From 0 to 10 minutes of hyperglycemic clamp
Second phase insulin/C-peptide response | From 10 to 60 minutes of hyperglycemic clamp
Area under the curve of insulin level during GLP-1 infusion under hyperglycemic clamp | From 60 minutes to 120 minutes during GLP-1 infusion under hyperglycemic clamp
Area under the curve of insulin/C-peptide level during GIP infusion under hyperglycemic clamp | From 120 minutes to 180 minutes during GIP infusion under hyperglycemic clamp
Difference of incretin sensitivity between diabetes patients and normal glucose tolerance subjects | From 60 minutes to 120 minutes during GLP-1 infusion under hyperglycemic clamp
  Area under the curve of C-peptide level during GLP-1 infusion under hyperglycemic clamp
Difference of first phase insulin/C-peptide response between diabetes patients and normal glucose tolerance subjects | From 0 to 10 minutes of hyperglycemic clamp
Difference of second phase insulin/C-peptide response between diabetes patients and normal glucose tolerance subjects | From 10 to 60 minutes of hyperglycemic clamp
Difference of area under the curve of insulin level during GLP-1 infusion under hyperglycemic clamp between diabetes patients and normal glucose tolerance subjects | From 60 minutes to 120 minutes during GLP-1 infusion under hyperglycemic clamp
Difference of Area under the curve of insulin/C-peptide level during GIP infusion under hyperglycemic clamp between diabetes patients and normal glucose tolerance subjects | From 120 minutes to 180 minutes during GIP infusion under hyperglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea